CLINICAL TRIAL: NCT03616548
Title: Surveillance of Allograft Rejection After Intestinal Transplantation Using a Magnifying Endoscopy With Narrow Band Imaging Scoring System ("VENCH" Score)
Brief Title: Surveillance of Allograft Rejection After Intestinal Transplantation Using Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: FEMH-105023-F
Record Dates: First submitted 2018-07-12; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Rejection of an Intestine Transplant
Keywords: intestinal transplantation; graft rejection; image enhanced endoscopy; narrow band imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intestinal transplantation (Other): Magnifying endoscopy under NBI system via chimney ileostomy after intestinal transplantation using a novel VENCH scoring system
  Interventions: Diagnostic Test: Endoscopic surveillance

INTERVENTIONS:
Diagnostic Test: Endoscopic surveillance — Magnifying endoscopy under narrow band imaging system via chimney ileostomy after intestinal transplantation

SUMMARY:
Intestinal failure (IF) which are characterized by inadequate maintenance of nutrition via normal intestinal function comprises a group of disorders with many different causes. If IF persists for more than a few days, it demands treatment with the intravenous supplement of water and nutrients, so-called parenteral nutrition (PN), to avoid life-threatening complications. However, PN dependency is associated with higher mortality and is therefore considered to have indications for intestine transplantation (IT). Graft acute cellular rejection is one of the most important reasons for graft failure. As a result, early identification of ACR and timely modification of anti-rejection medications has been considered to be associated with better graft and patient survivals. The diagnostic gold standard for ACR is mainly based on histology, but hours of delay by pathology may occur. Additionally, immunity in small bowel after transplantation should rely on a balance of innate and adaptive immune responses in the presence of the gut microbiota which the distribution may change after IT. Few researches investigated the association of changes of gut microbiota with graft rejection and narrow-band imaging endoscopy which can provide timely diagnosis of ACR in IT patients. In this study, we aimed to investigate the association of changes in mucosa-associated microbiota which was not addressed in the literature with rejection reaction by next-generation sequencing methods. We also use a new endoscopic scoring system to evaluate the diagnostic accuracy of rejection reaction using pathology as standard reference.

DETAILED DESCRIPTION:
Study design

This cohort study was conducted prospectively and approved by the ethics committee of Far Eastern Memorial Hospital (IRB No. FEMH-105023-F). Consecutive patients who received IT between November 2016 and September 2017 were enrolled. The inclusion criteria were as followings: post-IT patients older than 7-year-old, and with informed consent for endoscopy and biopsy. Those with bleeding tendency (platelet count <80k/ul, or prothrombin time international normalized ratio >1.5), without informed consent, or leukopenia (absolute neutrophil count <1,500/ul) were excluded.

Endoscopic and histological grading for allograft rejection Endoscopic surveillance was carried out after IT twice a week during the first month, once a week in the second month and then once per month until ileostomy closed. IEE examinations were performed with magnifying endoscopy (ME) which has powerful 80 times optical magnification under narrow-band imaging (NBI) system (Evis Lucera CLV-260NBI, GIF-H260Z endoscopy, Olympus Medical Systems Corp, Tokyo, Japan).14 ME was intubated through chimney ileostomy to anastomosis site to evaluate the changes of superficial mucosal surface and vascular architecture. Biopsy samples were taken from endoscopically suspicious rejection areas for histological examination. All the endoscopic procedures were done by one experienced endoscopist (C.S-C.) who was blinded to the histological reports.

All the histological reports were carried out by one experienced pathologist (C.C.-T.). The severity of histological rejection was graded according to followings:11 1) Indeterminate:

minimal histological changes including localized inflammatory infiltrate, crypt epithelial injury, increased crypt epithelial apoptosis but less than 6 apoptotic bodies/10crypts, no to minimal architectural distortion, no mucosal ulceration, or changes insufficient for the diagnosis of mild rejection; 2) Mild: mild localized inflammatory infiltrate with activated lymphocytes, mild crypt epithelial injury, increased crypt epithelial apoptosis > 6 apoptotic bodies/10crypts, mild architectural distortion but no mucosal ulceration; 3) Moderate: widely dispersed inflammatory infiltrate in lamina propria, diffuse crypt epithelial injury, increased crypt apoptosis with focal confluent apoptosis, more prominent architectural distortion, possible mild to moderate intimal arteritis, no mucosal ulceration; 4) Severe: features of moderate ACR, possible ulceration and denudation of mucosa, severe intimal arteritis or transmural arteritis may be seen. We classified those with apoptotic body≦1/10crypts and without other findings associated with indeterminate, mild, moderate to severe rejection as no rejection.

We used a novel endoscopic scoring system to record the architectural changes of microsurface and microvascularity of mucosa (Table 1). The observed endoscopic findings were recorded by the following five components ("V-E-N-C-H") graded 0 to 2 (Figure 1): 1) "V" (villi appearance): string-like (V-0), tongue-like (V-1), dome-like (V-2); 2) "E" (erythema of mucosa): no redness (E-0), sporadic (E-1), diffuse (E-2); 3) "N" (network of capillary): normal capillary loops (N-0), meandering caliber of capillary loops and loss of capillary loops in <50% villi under one maximal ME view (N-1), loss of capillary loops >50% villi under one maximal

ME view (N-2); 4) "C" (crypt widening): narrow (C-0), slightly widened within a width of one villi (C-1), markedly widened beyond a width of one villi (C-2); 5) "H" (heterogeneity of mucosal change): minimal (H-0), patch (H-1), diffuse (H-2).

Statistical analysis The continuous variables were expressed as mean ± standard deviation, whereas categorical variables were summarized as count (%). Pearson's correlation coefficient was used to analyze the severity of rejection between endoscopic scoring system and histological grading system. The significance levels were defined as p value <0.05 and the statistical analysis was performed using STATA software (version 11.0; Stata Corp, College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* Post-small intestinal transplantation patients
* Older than 7-year-old
* With informed consent for endoscopy and biopsy

Exclusion Criteria:

* Bleeding tendency (platelet count <80k/ul, PTINR >1.5)
* Without informed consent for endoscopy and biopsy
* Leukopenia (ANC <1,500/ul)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of endoscopic scoring system with severity of histological rejection | 1 year
  Endoscopists who are blinded to the clinical data recorded the imaging findings based on the V-E-N-C-H score, and the pathologists who are blinded to the clinical data reported the endoscopic biopsy specimen findings about rejection. Pearson's correlation test is used to evaluate the correlation between endoscopic and pathological findings.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Shuan Chung, MD, MSc, Study Director — Department of Internal Medicine, Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung CS, Tsai CC, Chen KC, Lin CK, Lee TH, Tsai HW, Chen Y. Surveillance of Rejection After Intestinal Transplantation Using an Image Enhanced Endoscopy "VENCH" Scoring System. Transplant Proc. 2021 Jan-Feb;53(1):364-370. doi: 10.1016/j.transproceed.2020.10.002. Epub 2020 Dec 9. PMID 33309060